CLINICAL TRIAL: NCT00940927
Title: Exclusion of Asthmatics From Clinical Trials Due to the 15 Percent Rule
Brief Title: Dose-response of Albuterol in Asthmatics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Kathryn Blake, Pharm.D., Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 93-41
Record Dates: First submitted 2008-06-27; First posted 2009-07-17 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: Albuterol; Forced expiratory volume in one second; Dose at fifty percent of maximum effect; Maximum effective dose; Metered dose inhaler; Nebulizer
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: albuterol — Albuterol administered sequentially 180mcg (MDI), 90mcg (MDI), 90mcg(MDI), 90mcg (MDI), 90mcg (MDI), 2.5mg (nebulized)
  Other Names: Proventil MDI; Proventil solution for nebulization

SUMMARY:
The purpose of this study was to determine the lung function response after increasing doses of albuterol (a bronchodilator) in children and adults with asthma.

DETAILED DESCRIPTION:
Inhaled short-acting b2-agonists (SABA) are the most potent bronchodilators used today to treat acute symptoms of asthma and albuterol, a partial b2-agonist, is the most frequently prescribed asthma medication in the US. Although universally used in for acute asthma symptoms, SABA have been associated with a significant degree of interpatient variability. Many studies have characterized the SABA dose to bronchodilator response relationship under controlled conditions. However, few studies have explored the magnitude and sources of bronchodilator response variability, and no studies have characterized the dose versus bronchodilator response relationship using population pharmacokinetic/pharmacodynamic (PPK/PD) modeling. In the present study, we characterized the relationship between inhaled doses of albuterol and bronchodilation in 81 children and adults with moderate to severe persistent asthma using a population pharmacodynamic approach. The purpose of this study was to obtain estimates of the pharmacodynamic parameters that characterize the dose-response curve, including maximal dose for bronchodilation, and to quantify and identify sources of interpatient pharmacodynamic variability.

ELIGIBILITY:
Eligibility Criteria:

* Well-defined history of physician diagnosed asthma
* Any ethnic background
* 8 to 65 years old
* Baseline pre-bronchodilator FEV1 of 40% to 80% predicted for age, height, and gender
* No oral corticosteroid use, emergency room visits, or hospitalizations within the previous 3 months
* Nonsmokers or less than a 5 pack-year history with no smoking in the previous year
* Normal physical exam and no confounding diseases were selected
* Able to withhold inhaled short-acting b2-agonists or inhaled anticholinergic drugs for 8 hours, oral antihistamines for 5 days, theophylline for 24 hours, and cromolyn, nedocromil, and inhaled corticosteroids for 2 hours prior to the study.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 1993-07; Primary Completion 1994-10 (Actual); Study Completion 1994-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn V Blake, Pharm.D., Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Result] Blake K, Madabushi R, Derendorf H, Lima J. Population pharmacodynamic model of bronchodilator response to inhaled albuterol in children and adults with asthma. Chest. 2008 Nov;134(5):981-989. doi: 10.1378/chest.07-2991. Epub 2008 Jun 26. PMID 18583517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from our asthma research clinic database or newspaper advertisements. Participants were recruited from 07/1993 to 10/1994.
Pre-assignment Details: Participants had to withhold inhaled short-acting beta2 agonist or inhaled anticholinergic drugs for 8 h, oral antihistamines for 5 days, theophylline for 24 h, and cromolyn, nedocromil, and inhaled corticosteroids for 2 h prior to the study.
Groups:
- Albuterol: Increasing doses of albuterol by MDI and nebulizer solution
Period: Overall Study
Arm/Group | Albuterol
Started | 81
Completed | 81
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Albuterol
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31
  Between 18 and 65 years | 48
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 81

OUTCOME MEASURES:

1. Primary Outcome: Effective Dose 50% (ED50)
Description: ED50 is the cumulative dose of albuterol required to bring about 50% of maximum effect of albuterol
Time Frame: 15 minutes after each dose
Measure: Number; unit: ug
Arm/Group | Albuterol
Number analyzed (Participants) | 81
ug | 141

2. Primary Outcome: Effect Maximum (Emax)
Description: Maximum percentage of predicted FEV1 effect
Time Frame: 15 minutes after each dose
Measure: Number; unit: percentage of predicted
Arm/Group | Albuterol
Number analyzed (Participants) | 81
percentage of predicted | 24.0

ADVERSE EVENTS:
Arm/Group | Albuterol
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No